CLINICAL TRIAL: NCT04959695
Title: Randomized Trial of Prolonged Exposure (PE) vs. PE With PE Coach Among Veterans With PTSD
Brief Title: Evaluation of the PE Coach Mobile Application Among Veterans With PTSD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Defense Centers of Excellence for Psychological Health and Traumatic Brain Injury (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D3503-R
Record Dates: First submitted 2021-05-03; First posted 2021-07-13 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Posttraumatic Stress Disorder
Keywords: posttraumatic stress disorder; prolonged exposure; exposure therapy; mobile applications; PE Coach; cognitive behavioral therapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Data analyst will be blind to the coding of assigned treatment intervention in the data set until analyses are complete.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Prolonged exposure with PE Coach (Experimental): The mobile application will be incorporated into each PE psychotherapy session and used to support homework between sessions.
  Interventions: Behavioral: PE Coach
- Prolonged exposure without PE Coach (Active Comparator): Standard PE treatment protocol without PE Coach
  Interventions: Behavioral: Prolonged exposure without PE Coach

INTERVENTIONS:
Behavioral: PE Coach — PE Coach is a treatment companion mobile application designed with features to support the tasks of prolonged exposure psychotherapy and the homework between sessions.
  Arms: Prolonged exposure with PE Coach
Behavioral: Prolonged exposure without PE Coach — Standard PE treatment protocol without PE Coach
  Arms: Prolonged exposure without PE Coach

SUMMARY:
Thousands of mental health mobile applications (apps) are available but limited research has been conducted on their effectiveness. VA has been a leader in mental health mobile app development and must research whether these apps work, and if so, how? PE Coach is a well-designed treatment companion app to one of the most researched, efficacious psychotherapies for PTSD (prolonged exposure), a treatment that has been broadly disseminated throughout VA mental health clinics. Research suggests that VA therapists find the app helpful in supporting patients. Preliminary results suggest that Veteran patients prefer to receive therapy with PE Coach and Veterans complete more recovery-oriented homework when they do. This study will randomize 124 Veterans with PTSD to treatment with or without PE Coach. The project will evaluate the effect of the app on PTSD-related functioning, quality of life, and PTSD symptoms. The investigators will test whether the app improves functioning and symptoms, increases homework, and reduces drop out.

DETAILED DESCRIPTION:
Veterans are at increased risk of posttraumatic stress disorder (PTSD), which negatively impacts social and occupational functioning and quality of life. Prolonged exposure (PE) is an evidence-based psychotherapy for PTSD that is effective in the treatment of Veterans. However, many Veterans drop out of psychotherapy for PTSD and many of those who complete PE still meet criteria for PTSD or do not achieve clinically meaningful change. The vast majority of Veterans with PTSD report neurobehavioral cognitive symptoms and may be at particular risk given that problems with executive functioning and prospective memory are related to PTSD treatment drop out and poorer treatment outcomes. The mechanisms of functioning and symptom change in PE include emotional activation during exposure, between-session habituation, and changes in PTSD-related negative cognitions. These mechanisms occur via verbally recounting and processing trauma memories (imaginal exposure) and approaching anxiety provoking situations in day-to-day life (in vivo exposure) and are achieved by daily homework exercises. Increased homework adherence predicts improved PTSD symptoms and functioning. To support patients participating in PE, the DoD/VA developed the mobile application (app) 'PE Coach'. The features of PE Coach were designed to enhance patients' ability to adhere with the homework critical to recovery. PE Coach may provide the cognitive and organizational support that Veterans with PTSD need to successfully complete treatment and maximize outcomes. However, little is known about the effectiveness of most mental health technology augmentations and this is true of PE Coach as well. Although the app is used in routine VA care and the VA recently invested in the software development required for an updated version of the app, no study has evaluated the impact of PE Coach on clinically relevant treatment outcomes. This study will conduct a randomized, controlled clinical trial to determine the efficacy of PE Coach and its impact on PTSD-related social and occupational functioning, PTSD symptoms, and homework adherence and dropout. The project will randomize 124 Veterans with PTSD to either PE +PE Coach or Usual PE (without PE Coach). Participants in both conditions will have identical homework activities assigned, but those with PE + PE Coach will receive all of their homework activities through the PE Coach app, while those in Usual PE will receive their homework through separate, standard workbook handouts and digital audio recording device. Veterans will participate in 8-15 weekly individual PE psychotherapy sessions, based on defined termination criteria and delivered consistent with the published treatment manual. Outcome assessments will be conducted at baseline, half-way through treatment, post-treatment, and at 1- and 4- month follow-ups. The primary outcome measure will be the Posttraumatic Stress Related Functioning Inventory (PRFI). PTSD symptoms will be assessed using the gold-standard Clinician Administered PTSD Scale for DSM-5, Revised which will be conducted by independent assessors blind to treatment condition. Functioning, quality of life, self-reported PTSD, and depression will be monitored every-other PE session, throughout treatment. An external PE expert will code 15% of PE sessions to monitor the fidelity of psychotherapy to the treatment protocol, and homework adherence will be reported at each session to test the impact of PE Coach on adherence. VA has been a leader in mental health mobile app development and must respond to the call for research on whether these apps work, and if so, how? This study addresses that need by testing the efficacy of PE Coach, a treatment companion to one of the most researched, efficacious psychotherapies for PTSD, and a treatment that has been broadly disseminated throughout VA mental health clinics. Results can help inform whether VA should invest in systematic implementation and dissemination of PE Coach as a routine part of PE training in VA.

ELIGIBILITY:
Inclusion Criteria:

* Veterans aged 18-65
* enrolled in VA healthcare and eligible for VA PTSD psychotherapy
* current diagnosis of PTSD based on CAPS-5, Minimum total severity score of 26 or higher
* English language fluency
* willingness to participate in individual, in-person or telemental health PE psychotherapy including use of a mobile device

Exclusion Criteria:

* neurological conditions (based on review of the volunteer's medical record) that are severe enough to interfere with PE treatment and assessments (i.e., diagnosed Major Neurocognitive Disorder, severe neurological disorders (e.g., ALS), and those with severe TBI history). Neurological disorders that may result in mildly impaired cognitive function (such as multiple sclerosis or those with history of mild or moderate severity TBI) will be eligible, pending a score of 6 or higher on the Short Portable Mental Status Questionnaire
* current intent to suicide
* behavioral patient record flag in the VA medical record
* a history of a serious mental health condition listed in their medical record problem list that is known to include psychotic symptoms, such as schizophrenia or a depressive disorder with psychotic features. We will also ask for self -reported indicators of psychosis, using an existing interview template
* in an ongoing threatening situation (e.g. domestic violence)
* positive screen for severe alcohol use disorder, as indicated by an AUDIT score equal to or higher than 13 or 15 for women and men, respectively
* prior history of 3 or more sessions of PE therapy for PTSD
* other current psychotherapy for PTSD that is recommended (with at least weak strength) in the VA/DoD Clinical Practice Guideline for the treatment of PTSD
* a physical condition that interferes with the proper use of a mobile device.
* not stable on psychotropic medications for at least 6 weeks prior to enrollment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2022-07-29 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in Posttraumatic Stress Related Functioning Inventory (PRFI) from baseline to mid-treatment, post-treatment, 1-month post-treatment f/up, 4-month post-treatment f/up | Pre-treatment (Baseline), approx week 8 (mid-treatment), approx. week 16 (post-treatment), approx week 20 (1-month f/up), approx week 32 (4-month f/up)
  The PRFI is a 33-item, self -report measure of,functioning related to three domains: work and school, relationships, and lifestyle. Each domain is assessed with two subscales, including a Symptom Cluster Impact scale, which assess the impact of each DSM-5 PTSD symptom cluster on functioning in that domain, and a Total Symptom Impact subscale, which assesses the impact of all PTSD symptoms.

SECONDARY OUTCOMES:
Change in World Health Organization Disability Assessment Schedule 2.0 (WHODAS 2.0) from baseline to mid-treatment, post-treatment, 1-month post-treatment f/up, and 4-month post-treatment f/up | Pre-treatment (Baseline), approx week 8 (mid-treatment), approx. week 16 (post-treatment), approx week 20 (1-month f/up), approx week 32 (4-month f/up)
  The WHODAS 2.0 is a 36-item self -report measure that assesses disability in the past 30 days related to general medical and psychiatric disorders across six domains of functioning (cognition, mobility, self -care, getting along, life activities, participation) and provides subscale scores and an overall disability score ranting from 0 (no disability) to 100 (full disability).
Change in World Health Organization Quality of Life Instrument, Abbreviated Version (WHOQOL-BREF) from baseline to mid-treatment, post-treatment, 1-month post-treatment f/up, and 4-month post-treatment f/up | Pre-treatment (Baseline), approx week 8 (mid-treatment), approx. week 16 (post-treatment), approx week 20 (1-month f/up), approx week 32 (4-month f/up)
  The WHOQOL-BREF is a well-validated, 26-item self -report measure that assesses quality of life across four domains: physical health, psychological, social relationship, and environment. Patients report on a 5-point Likert scale their experience/satisfaction across various life domains over the prior two weeks.
Change in Clinical Global Impression of Change - Symptoms and Improvement (CGI-Symptoms) from mid-treatment to post-treatment, 1-month post-treatment f/up, and 4-month post-treatment f/up | approx week 8 (mid-treatment), approx. week 16 (post-treatment), approx week 20 (1-month f/up), approx week 32 (4-month f/up)
  CGI-Symptoms will be measured using a 7-point Likert scale asking participants (at post-treatment and at f/u) to rate their perception of change in PTSD symptoms as a result of treatment as "very much improved," 2 or "much improved," 3 or "minimally improved," 4 or "no change," 5 or "slightly worse," 6 or "much worse," and 7 or "very much worse" . The same scale/anchors will be used to have patients rate any change in their ability to "participate meaningfully in life activities" (Improvement).
Change in Beck Depression Inventory-II (BDI-II) from baseline to mid-treatment, post-treatment, 1-month post-treatment f/up, 4-month post-treatment f/up | Pre-treatment (Baseline), approx week 8 (mid-treatment), approx. week 16 (post-treatment), approx week 20 (1-month f/up), approx week 32 (4-month f/up)
  The BDI-II is a 21-item self -report measure of the severity of depressive symptoms. Patients rate each item using a 4-point Likert-type scale ranging from 0 (least severe) to 3 (most severe). Ratings are summed to yield a total severity score, in which higher scores indicate higher levels of depressive symptoms.
Change in Columbia-Suicide Severity Rating Scale (C-SSRS) from baseline to mid-treatment, post-treatment, 1-month post-treatment f/up, and 4-month post-treatment f/up | Pre-treatment (Baseline), approx week 8 (mid-treatment), approx. week 16 (post-treatment), approx week 20 (1-month f/up), approx week 32 (4-month f/up)
  The C-SSRS is a gold-standard, clinician assessment of suicidal ideation and suicidal behavior. The C-SSRS measures four separate constructs: severity of ideation, intensity of ideation, behavior, and lethality. The patient is rated by the assessor as to the experience of the highest level experienced of each construct over the specified period.
Change in PTSD Checklist for DSM-5 (PCL-5) from baseline to mid-treatment, post-treatment, 1-month post-treatment f/up, 4-month post-treatment f/up, and every other approximately weekly treatment session | Pre-treatment (Baseline), approx week 8 (mid-treatment), approx. week 16 (post-treatment), approx week 20 (1-month f/up), approx week 32 (4-month f/up)
  The PCL-5 is a widely used and well-validated self -report measure of PTSD symptoms, and comprises 20 items corresponding to each of the DSM-5 symptom criteria for PTSD. The PCL-5 assesses the patient's experience of symptoms over the past month, or week, and each item is rated on how bothersome the patient has found that particular symptom (0 = not at all; 1 = a little bit; 2 = moderately; 3 = quite a bit; 4 = extremely). Thus, scores on the PCL-5 range from 0-80, with higher scores indicating more severe PTSD symptoms.
Sum of Utility of Techniques Inventory (UTI) at each weekly treatment session starting treatment session 2 | Weekly treatment Sessions 2-15 (approx weeks 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16)
  The UTI is a self -report measure that asks patients to retrospectively report the frequency and perceived helpfulness of assigned PE homework. Frequency of homework adherence is rated from 0 (not at all) to 5 (more than 10 times). Perceived helpfulness responses range from 1 (not helpful at all) to 5 (extremely helpful).
PE Homework Daily Diary | Weekly treatment Sessions 2-15 (approx weeks 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16)
  A calendar documenting the raw count of days of self-reported adherence to assigned imaginal and in vivo homework (typically, 0-7 for each) in the week prior to each PE session.
Change in Neurobehavioral Symptom Inventory from baseline to mid-treatment, post-treatment, 1-month post-treatment f/up, 4-month post-treatment f/up | Pre-treatment (Baseline), approx week 8 (mid-treatment), approx. week 16 (post-treatment), approx week 20 (1-month f/up), approx week 32 (4-month f/up)
  The NSI is a 22-item, self-report measure of neurobehavioral symptoms that includes four symptom clusters: Cognitive, Somatosensory, Affective, and Vestibular.
Change in Posttraumatic Stress Related Functioning Inventory (PRFI) across treatment, measured every other treatment session | Session 2 (approx week 3), Session 4 (approx week 5), Session 6 (approx week 7), Session 8 (approx week 9), Session 10 (approx week 11), Session 12 (approx week 13), Session 14 (approx week 15)
  The PRFI is a 33-item, self -report measure of functioning related to three domains: work and school, relationships, and lifestyle. Each domain is assessed with two subscales, including a Symptom Cluster Impact scale, which assess the impact of each DSM-5 PTSD symptom cluster on functioning in that domain, and a Total Symptom Impact subscale, which assesses the impact of all PTSD symptoms.
Change in Beck Depression Inventory-II (BDI-II) across treatment, measured every other treatment session | Session 2 (approx week 3), Session 4 (approx week 5), Session 6 (approx week 7), Session 8 (approx week 9), Session 10 (approx week 11), Session 12 (approx week 13), Session 14 (approx week 15)
  The BDI-II is a 21-item self -report measure of the severity of depressive symptoms. Patients rate each item using a 4-point Likert-type scale ranging from 0 (least severe) to 3 (most severe). Ratings are summed to yield a total severity score, in which higher scores indicate higher levels of depressive symptoms.
Change in PTSD Checklist for DSM-5 (PCL-5) across treatment, measured every other treatment session | Session 2 (approx week 3), Session 4 (approx week 5), Session 6 (approx week 7), Session 8 (approx week 9), Session 10 (approx week 11), Session 12 (approx week 13), Session 14 (approx week 15)
  The PCL-5 is a widely used and well-validated self -report measure of PTSD symptoms, and comprises 20 items corresponding to each of the DSM-5 symptom criteria for PTSD. The PCL-5 assesses the patient's experience of symptoms over the past month, or week, and each item is rated on how bothersome the patient has found that particular symptom (0 = not at all; 1 = a little bit; 2 = moderately; 3 = quite a bit; 4 = extremely). Thus, scores on the PCL-5 range from 0-80, with higher scores indicating more severe PTSD symptoms.
Change in Clinician Administered PTSD Scale for DSM-5, Revised (CAPS-5-R) from baseline to mid-treatment, post-treatment, 1-month post-treatment f/up, and 4-month post-treatment f/up | Pre-treatment (Baseline), approx week 8 (mid-treatment), approx. week 16 (post-treatment), approx week 20 (1-month f/up), approx week 32 (4-month f/up)
  The CAPS-5-R is a recent revision of the CAPS-5. CAPS-5-R assesses for the frequency and intensity of DSM-5 symptoms. Frequency is assessed per the patient report (e.g, times per month or percentage of the time the symptom is present). Intensity of symptoms is scored as absent, minimal, clearly present, pronounced, and extreme. Two intermediate intensity ratings are available for clearly present/pronounced, and pronounced/extreme. The combination of frequency and intensity ratings determine the 0 to 10 severity score for each item. Although the range for item severity scores has expanded from 0-4 on the CAPS-5 to 0-10 on the CAPS-5-R, CAPS-5 scores are nested in the CAPS-5-R scoring grid, so either scoring method can be used. Although we will administer the CAPS-5-R, we will use CAPS-5 scoring for the inclusion criterion.

CONTACTS AND LOCATIONS:
Overall Officials: Greg M. Reger, PhD, Principal Investigator — VA Puget Sound Health Care System Seattle Division, Seattle, WA
Locations (1):
- VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
The data sets include research involving human subjects. A de-identified, anonymized dataset will be created and shared. Subject to IRB approval, de-identified data will be released to a local VAPSHCS and/or national VA research data repository for release to non-VA protocols. The VA research data repository administrator will be responsible for reviewing and responding to requests to release data to non-VA requestors. A data use agreement compliant with VHA Handbooks 1200.12 and 1605.1 will be required between VHA and the requestor. Review and approval by VA privacy officer is required prior to disclosure.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available after release to a local or national VA research data repository and subsequent to all required approvals. Data will be de-identified as required by VHA Hbk 1605.1, Appendix B. All 18 HIPAA identifiers will be removed from the data, including any unique study identifier(s). If random number assigned to de-identified data set, VA will not retain crosswalk, link or other method to re-identify subjects. Proprietary information to be excluded. Subject to IRB approval, data released to VA research data repository. DUA prohibits requestor from re-identifying subjects. Privacy office approval required.
Access Criteria: The VA research data repository administrator will be responsible for reviewing and responding to requests to release data to non-VA requestors. A data use agreement compliant with VHA Handbooks 1200.12 and 1605.1 will be required between VHA and the requestor. Review and approval by VA privacy officer is required prior to disclosure.

REFERENCES:
- [Derived] Reger GM, Smolenski D, Williams R, Norr AM, Foa E, Kuhn E, Schnurr PP, Weathers F, Zoellner L. Design and methods of a randomized controlled trial evaluating the effects of the PE Coach mobile application on prolonged exposure among veterans with PTSD. Contemp Clin Trials. 2023 Apr;127:107115. doi: 10.1016/j.cct.2023.107115. Epub 2023 Feb 8. PMID 36758935